CLINICAL TRIAL: NCT05280899
Title: The Impact of Varying Weightbearing Restrictions on Postoperative Outcomes Following Arthroscopic Surgery for Femoroacetabular Impingement: a Randomized Trial
Brief Title: Weightbearing Restrictions on Postoperative Outcomes Following Arthroscopic Surgery for FAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hip WB RCT
Record Dates: First submitted 2021-12-14; First posted 2022-03-15 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Femoro Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Weight-Bearing; Partial Weight-Bearing

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded trial will be completed with patients receiving one of two differing post-operative weightbearing recommendations
Who Masked: Outcomes Assessor
Masking Description: Patients and surgeons will not be blinded to group allocation (weight-bearing status). The study Research Coordinator will perform randomization therefore they will also not be blinded to group allocation. The assessor for the functional and return to sport outcomes will be blinded to group allocation. To protect blinding, before each functional testing appointment, the blinded tester will remind patients not to reveal their group (weightbearing status).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Weight-bearing (PWB) (Active Comparator): Patients will PWB for 3 weeks following surgery, followed by a gradual return to FWB.
  Interventions: Other: Partial Weight-bearing
- Weight-bearing As Tolerated (WBAT) (Experimental): Patients will WBAT immediately following surgery.
  Interventions: Other: Weight-bearing As Tolerated

INTERVENTIONS:
Other: Weight-bearing As Tolerated — The WBAT group will be instructed to bear weight as tolerated immediately following their surgical procedure. The rehabilitation protocols provided will be identical beyond the initial weightbearing recommendations. Following the initial protection phase (three weeks), whereby the two weightbearing interventions will be provided, patients will progress through standardized phases including mobility and neuromuscular retraining, muscle balance and strengthening, functional training, and finally, advanced training for return to work and sport.
  Arms: Weight-bearing As Tolerated (WBAT)
Other: Partial Weight-bearing — The PWB group will be instructed to bear weight to a maximum of 20 lbs of bodyweight on the operative limb for the initial three weeks (termed "toe touch"), with graduated return to full weightbearing thereafter.
  Arms: Partial Weight-bearing (PWB)

SUMMARY:
The purpose of this single-blinded (assessor) randomized trial is to compare patient-reported, clinical and functional outcomes in patients randomized to weight-bearing as tolerated (WBAT) or partial weight-bearing (PWB) restrictions following arthroscopic surgery for femoroacetabular impingement (FAI) up to 12-months postoperative.

DETAILED DESCRIPTION:
The purpose of this single-blinded (assessor) randomized trial is to compare patient-reported, clinical and functional outcomes in patients randomized to weight-bearing as tolerated (WBAT) or partial weight-bearing (PWB) restrictions following arthroscopic surgery for femoroacetabular impingement (FAI) up to 12-months postoperative. The primary objective is to compare the effects of WBAT or PWB restrictions on PROMS (International Hip Outcome Tool (iHOT33)) and clinical measures following arthroscopic intervention for FAI up to one-year post-operative. The secondary objective will be to assess differences in return to sport (RTS) PROMS, functional performance, and lower extremity kinetics, kinematics, and muscle activity during in patients randomized to either WBAT or PWB at six- and 12-months post-operative. The goal will be to answer if there are differences between a WBAT versus PWB rehabilitation protocol on patient-reported quality of life as measured by the International Hip Outcome Tool (iHOT33) at 12-m post-operative for patients undergoing primary hip arthroscopy for the treatment of FAI.

ELIGIBILITY:
Inclusion Criteria:

* 16 - 50 years of age at time of surgery
* Diagnosis of FAI (cam, pincer, mixed) based on the 2016 Warwick Agreement. All 3 criteria below must be met:

  1. Symptoms of motion- or position-related pain in the hip or groin
  2. Clinical signs consistent with FAI such as: decreased hip flexion and internal rotation, or positive impingement sign
  3. Radiographic evidence (on BOTH x-ray AND non-contrast MRI) of intra-articular pathology consistent with FAI as determined by the treating surgeon.
* Failed conservative interventions of at least 3 months (i.e. physiotherapy)
* Have symptom relief with intra-articular injection of local anaesthetic
* Unilateral or bilateral surgical intervention (note: unilateral required to ensure the weight bearing guidelines are followed)
* Are willing to be followed for 12 months post-operative.

Eligibility for 'return to sport' cohort:

Additional assessment measures related to return to sport will be collected on the patient who meet the following criteria:

* are or were previously actively involved in sport as indicated by a pre-operative Hip Sports Activity Scale score of four of greater
* indicate a post-operative goal to return to sport following their procedure

Exclusion Criteria:

Clinical:

* Previous surgery on the affected hip, or other major lower extremity orthopaedic surgery
* Active joint or systemic infection, significant muscle paralysis, significant lower extremity or medical comorbidity that could alter the effectiveness of the surgical intervention (e.g. polymyalgia rheumatica)
* Unable to speak or read English/French
* Unable or unwilling to be followed for 1 year or complete functional testing
* Presence of chronic pain syndromes
* History of pediatric hip disease (i.e. Slipped Capital Femoral Epiphysis, Legg-Calve-Perthes Disease)
* Ongoing litigation or compensation claims related to the hip (including Workers' Compensation)

Radiographic:

* Osteoarthritis greater than Tönnis Grade 1 on affected hip
* Lateral central edge angle <19°
* Dysplasia in patients with broken Shenton line (i.e. Severe acetabular deformity present)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool (iHOT-33) | 12 months
  The iHOT uses 33 questions to measure health-related quality of life. It is the primary outcome and has been validated for use in this population. Questions are evaluated on a 100-point visual analog scale (VAS) response format, where "0" represents the worst possible quality of life, and "100" represents the the best.

SECONDARY OUTCOMES:
Non-contrast MRI | 0 months
  Non-contrast MRI will be documented and used to assess for the presence of a labrum tear, articular cartilage lesions, cystic changes within the femoral neck or acetabulum.
Computed Tomography (CT) Scan | 0 months
  All patients will undergo a pre-operative CT scan with three dimensional reconstructions of the hip joint. This permits improved visualization of the boney impingement lesions that are being treated at the time of surgery.
The Copenhagen Hip and Groin Outcome Score (HAGOS) | 12 months
  HAGOS includes six separate subscales assessing pain, symptoms, physical function in daily living, physical function in sport and recreation, participation in physical activity and hip/groin-related quality of life and is designed for use with young to middle-aged physically active individuals with hip pain. Questions are answered on a five-point scale, with "0" indicating no problems, and 4 indicating extreme problems.
Hip Sports Activity Scale (HSAS) | 12 months
  HSAS will indicate the patient's pre surgical and current level of sports participation using a nine-point scale ranging from no recreational or competitive sports ("0") to competitive, elite level sport ("8").
Hip Return to Sport after Injury scale (Hip-RSI) | 12 months
  The Hip-RSI includes six questions regarding an athlete's readiness to return to sport using questions evaluating the athlete's emotional state, their confidence in performance, and their appraisal of risk related to their sport and injury. Each question is graded from 0 to 100, with variable definitions including 0 being "Not confident at all", and 100 being "fully confident", with higher scores indicating higher readiness to return to sport.
Single Assessment Numeric Evaluation (SANE) score | 12 months
  The SANE score is a single question that asks patients to rate their affected hip as a percentage of normal to provide a simple and efficient measure of patient outcome 8. All patients will be asked the following question during their clinical exam: "How would you rate your affected hip today as a percentage of normal (0% to 100% scale with 100% being normal)?"
Rate of surgical complications, re-operations and revision surgeries | 12 months
  Surgical complications will be documented at the time of surgery and at each postoperative interval. A surgical complication is defined as any undesirable, unintended and direct result of an operation affecting the patient that would not have occurred had the operation gone well as could reasonably be hoped (i.e. infection, neurological injury). Revisions and re-operations will be documented, including the reason for failure, date of revision/reoperation, and the procedure performed. A revision is defined as a subsequent surgery performed to correct or compensate for the initial procedure. Re-operation is defined as any surgical procedure other than a revision.
Postoperative Pain and Medication | 14 days
  Postoperative pain will be self-reported on a 100mm visual analogue scale (VAS) in a logbook. Medication type and quantity will also be documented. The Postoperative Pain and Medication Logbook has been previously used by the authors in an ACL population. ) on the scale will represent "No pain at all", and 100 will represent "Wort pain possible".
Hip Isometric Muscle Strength | 12 months
  Isometric hip abduction and extension will be measured in the side-lying and prone positions with a hand-held dynamometer (Chatillon DFX2, Ametek, PA, USA) positioned 5 cm proximal to the most prominent aspect of the malleolus. Four maximal holds of 5 seconds separated by 15 seconds rest will be completed after two submaximal familiarizations with 30 seconds of rest between attempts 25.
Hip Isokinetic Muscle Strength | 12 months
  Five repetitions of concentric, isokinetic hip flexion and extension peak torque will be measured on an isokinetic dynamometer (Biodex, Medical System 3, NY, USA) with the patient in the supine position (0 degrees to 50 degrees hip flexion at 60 degrees/second). Hamstring strength will be measured with the NordBord Hamstring Dynamometer (Vald, Qld, Aus).
Jump Testing | 12 months
  Participants will complete a standardized battery consisting of the drop vertical jump (jumping from a 30cm box to force plates positioned at a distance of 50% of their height from the starting line), a counter movement jump (jumping from the standing position with the hands on the hips on dual force plates), a squat jump and a single leg countermovement jump. Jump attempts will be recorded with three cameras (one frontal, two sagittal plane views) to assess maximal joint angles of the ankle, knee and hip. Anatomical markers for kinematic analysis of the lower extremity will be placed bilaterally at the following sites: anterior superior iliac spine, lateral iliac crest, greater trochanter, mid-thigh, medial and lateral knee joint line, tibial tubercle, mid-shank, distal shank, medial and lateral malleolus, and to the foot at the heel, dorsal surface of the lateral mid-foot, and toe with adhesive tape to the shoes
Hop Tests | 12 months
  A standardized battery of hop tests will be completed including the single leg hop, triple hop, triple crossover hop and medial and lateral triple hops for distance. Distances will be measured from the starting line to the posterior surface of the heel at landing with a standard tape measure
5-0-5 Change of Direction (505) | 12 months
  The participant will run 15 m, complete an 180o change of direction and run back to the starting line, with timing gates positioned at the 10 m mark to time the direction change (Brower Timing Systems, UT, USA).
Electromyography of the gluteal muscles | 12 months
  Electromyographic (EMG) data will be collected per Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM) standards on the upper and lower portions of the gluteus maximus muscle group (two finger widths above and below the midline between the posterior superior iliac spine and the greater trochanter of the femur for the upper and lower gluteus maximum respectively) and gluteus medius (proximal 1/3 of the distance between the iliac crest and the greater trochanter) following preparation of the skin (shaving and cleaning of the skin with isopropyl alcohol). Prior to testing, maximal voluntary isometric contractions of the gluteal muscles will be completed for normalization purposes. Peak EMG amplitudes for the gluteal muscles normalized to maximal voluntary isometric contractions will be collected during isometric hip abduction and extension and isokinetic hip flexion and extension and compared between the affected and unaffected limb, and between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Devin Lemmex, MD, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No